CLINICAL TRIAL: NCT06621329
Title: Transnasal Sphenopalatine Ganglion Block for Treatment of Acute Subarachnoid Hemorrhage Associated Headache
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Agnes Marshall Walker Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2160233
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: SAH (Subarachnoid Hemorrhage); Headache
Keywords: aSAH; peripheral nerve block; sphenopalatine ganglion; subarachnoid hemorrhage; headache
MeSH Terms: conditions — Subarachnoid Hemorrhage; Headache

STUDY DESIGN:
Intervention Model Description: Both arms will receive standard of care medications for headache management. The intervention group will receive an SPG block at a specific threshold defined in the study protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard of Care Medications for Headache (No Intervention): Control arm participants will receive standard of care medications, as defined in a headache protocol, to treat subarachnoid associated headache.
- Transnasal SPG Block and Standard of Care Medications (Experimental): Intervention arm participants will receive standard of care medications, as defined in a headache protocol, with the addition of transnasal SPG blocks when a predefined threshold is met per the study protocol.
  Interventions: Combination Product: Transnasal sphenopalatine ganglion block

INTERVENTIONS:
Combination Product: Transnasal sphenopalatine ganglion block — Transnasal sphenopalatine ganglion blocks will be performed using the Tx360 device. Medications used during the procedure include 0.75% bupivacaine with or without 1 mg of preservative free dexamethasone.
  Other Names: SPG block; peripheral nerve block
  Arms: Transnasal SPG Block and Standard of Care Medications

SUMMARY:
The study titled "Transnasal sphenopalatine ganglion block for treatment of acute subarachnoid hemorrhage associated headache" is a randomized controlled pilot study aimed at evaluating the efficacy of a transnasal sphenopalatine ganglion (SPG) block in addition to standard pain medication for reducing headache severity in patients with acute subarachnoid hemorrhage (aSAH). The study also examines whether this intervention can reduce opioid requirements during hospitalization and upon discharge.

DETAILED DESCRIPTION:
The study is designed to test the hypothesis that the addition of a transnasal SPG block to standard pain medication is more effective than medication alone in reducing headache associated with acute subarachnoid hemorrhage. It involves 40 participants who meet specific inclusion criteria, such as being over 18 years old, having a secured aneurysm, and the ability to verbalize pain scores. Those with conditions like recent nasal or facial trauma, allergies to specific anesthetics, or pregnancy are excluded.

Participants are randomized into two groups: one receiving the standard care medication for headache and the other receiving both the standard care and a transnasal SPG block. The SPG block is administered using a needleless device called the Tx360, which allows for the medication to be instilled directly to the the sphenopalatine ganglion via the nasal passageways.

Data on pain scores and opioid usage are collected and analyzed using statistical methods to assess the effectiveness of the SPG block. The study also includes safety monitoring to track any adverse effects from the intervention. The entire study spans approximately 24 months, with individual participation lasting up to four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Acute subarachnoid hemorrhage
* Age greater than 18 years
* Secured aneurysm
* Patient can verbalize pain score to clinician, nurse, medical translator, or surrogate decision
* maker
* Patient or surrogate decision maker is available to consent

Exclusion Criteria:

* Less than 18 years old
* Unsecured aneurysm
* Pregnant or lactating
* Prisoner
* Unable to verbalize pain score to clinician, nurse, medical translator, or surrogate decision maker
* Nasal or facial trauma or surgery within the last three months
* Allergy to lidocaine, bupivacaine, or dexamethasone
* Patient is unable to consent and no available surrogate decision maker

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Numerical pain rating scale | From enrollment until ICU discharge, up to 14 days
  Pain scores will be obtained at regular intervals to compare pain control between the two arms. Pain scores will be collected multiple times throughout each ICU day, up to ICU day 14.

SECONDARY OUTCOMES:
Morphine milligram equivalents (MME) | From enrollment to hospital discharge, up to 14 days
  Total Morphine milligram equivalents per ICU day will be collected for up to 14 days. Total morphine milligram equivalents will also be collected on the day of hospital discharge. Total morphine milligram equivalents for ICU course and total morphine milligram equivalents on day of discharge will be compared between the two arms.

OTHER OUTCOMES:
Vasospasm | From enrollment to ICU discharge, up to 14 days
  Incidence of vasospasm during ICU course will be collected for both arms.
Incidence of adverse events related to SPG block procedure | From enrollment to hospital discharge, up to 14 days
  Adverse reactions or events related to the SPG block procedure will be tracked and documented.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Picinich, MS, AGACNP-BC, CCRN, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Undecided